CLINICAL TRIAL: NCT05307809
Title: Cytokine Expression in Sera, Ex Vivo Stimulated Peripheral Blood Mononuclear Cells Culture, and Skin in Psoriasis - Comparison of Patients with and Without Joint Involvement
Brief Title: Cytokine Expression in Psoriasis Patients with and Without Joint Involvement
Acronym: CYNEPSA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CYNEPSA
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Psoriasis; Psoriatic Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Psoriasis (Experimental)
  Interventions: Other: Blood sample collection; Other: Skin sample collection
- Psoriatic arthritis (Experimental)
  Interventions: Other: Blood sample collection; Other: Skin sample collection
- Controls (Active Comparator)
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — Blood sample collection
Other: Skin sample collection — Skin sample collection
  Arms: Psoriasis; Psoriatic arthritis

SUMMARY:
The objective of the resarch is to study the cytokine profile of patients with psoriatic arthritis and psoriasis in order to better understand the pathophysiology of the disease and the contribution of cytokines to the presence or absence of joint involvement. This research will compare cytokines levels in sera, in PBMC culture after LPS or CD3/CD28 agonist antibodies, and in skin biopsy.

DETAILED DESCRIPTION:
Psoriatic arthritis and Cutaneous Psoriasis are polygenic inflammatory disorders with high burden on the quality of life of patients. Pathophysiology of those disease remain incompletely understood. Recent publications seem to demonstrate an implication of IL-1 family cytokines in the pathogenesis of both diseases. In the literature, results are discordant and focus mainly on cytokines levels in serum of patients. Moreover, few studies compare psoriatic arthritis patients with cutaneous psoriasis patients. We propose here to study cytokines profiles of patients with those conditions in sera, after ex-vivo stimulation of peripheral blood mononuclear cells, and in skin biopsies.

ELIGIBILITY:
Inclusion criteria:

* For psoriasis patients :

  * Age over 18 years old
  * Signed informed consent
  * 5 year old psoriasis at least
  * At least one skin lesion over 2 cm
  * Without any articular symptoms
  * Without any DMARDs
  * Without anticoagulant treatments or coagulation disease
  * With normal articular and enthesis sonography
* For psoriatic arthritis patients :

  * Age over 18 years old
  * Signed informed consent
  * Psoriatic arthritis according to CASPAR criteria
  * Without any DMARDs
  * Without anticoagulant treatments or coagulation disease
  * With at least one synovitis at inclusion
* For controls

  * Age and sex matched with a patient without any rheumatic or dermatologic medical conditions
  * No treatment with corticosteroïds or non-steroïdial anti-inflammatory drugsAge over 18 years old

Exclusion criteria:

▪ For psoriasis patients :

* Joint damage according to CASPAR criteria
* Echography activity in favor of chronic inflammatory rheumatism
* For patients and controls:
* Without social protection rights
* People under judiciary protection, of less than 18 years old, pregnant woman, breast feeding women, jailed patients.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2026-08-17 (Estimated); Study Completion 2026-08-18 (Estimated)

PRIMARY OUTCOMES:
Comparison of cytokine levels in sera, after culture of PBMC stimulated with LPS or CD3/CD28 agonist antibodies between the three groups | At inclusion
  Comparison of cytokine levels in sera, after culture of PBMC stimulated with LPS or CD3/CD28 agonist antibodies between the three groups

SECONDARY OUTCOMES:
Comparison of cytokine levels in skin biopsies between Psoriatic Arthritis and Cutaneous Psoriasis patients | At inclusion
  Comparison of cytokine levels in skin biopsies between Psoriatic Arthritis and Cutaneous Psoriasis patients
Correlation of cytokine levels with rheumatologic disease activity, or dermatologic disease activity | At inclusion
  Correlation of cytokine levels with rheumatologic disease activity, or dermatologic disease activity

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LARID, Principal Investigator — Poitiers University Hospital
Locations (1):
- Chu Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Yes
Publication of the results
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Results will be published in a scientific journal
Access Criteria: Upon reasonable request to authors after article publication